CLINICAL TRIAL: NCT01546285
Title: B40 Non-Invasive Blood Pressure Equivalency Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 118.04-2011-GES-0002
Record Dates: First submitted 2012-02-28; First posted 2012-03-07 (Estimated); Results first posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-05

CONDITIONS: Blood Pressure
Keywords: The focus of this study is to demonstrate that DINAMAP® SuperSTATTM NIBP algorithm has been implemented correctly without performance losses to the B40 monitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood Pressure Reading (Experimental): Simultaneous blood pressure readings with DINAMAP PRO1000 and B40 monitor; total of 6 successful readings
  Interventions: Device: Blood Pressure Readings on B40 Patient Monitor

INTERVENTIONS:
Device: Blood Pressure Readings on B40 Patient Monitor — Simultaneous blood pressure reading on the Investigational B40 patient monitor and DINAMAP PRO1000 patient monitor

SUMMARY:
The purpose of this study is to demonstrate equivalency of the GE Healthcare B40 Patient Monitor noninvasive blood pressure (NIBP) parameter compared to the reference device.

DETAILED DESCRIPTION:
Automated non-invasive blood pressure devices have a long history. These devices first made their appearance in the mid-1970's. Since that time, there have been many improvements in the performance of these devices. Specifically, when making changes to the algorithms that control these devices, the goals are: to improve accuracy and precision in the blood pressure (BP) estimates, to reduce the time needed to determine the BP estimates, to increase comfort for the patient, and to work through artifacts and arrhythmias that are often present in the clinical environment.

The purpose of this study is to demonstrate equivalency of the GE Healthcare B40 Patient Monitor noninvasive blood pressure (NIBP) parameter compared to the reference device.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent or have a legally authorized representative including a parent or guardian provide written informed consent
* Within the age range from older than 3 years old to 75 years old (adult and child)
* Ability to maintain proper placement of cuff and/or probe and/or sensor

Exclusion Criteria:

* Neonates (ages 0-29 days) and infants (30 days to 3 years old) shall be excluded
* Any subject deemed too unstable, by clinician's discretion, or for another reason deemed unacceptable for study by the clinician
* Known dysrhythmias (when applicable)
* Known disease state that compromises circulation to the extremity
* Vigorous exercise prior to participating in the study
* Excessive movement or excitability causing false values or no determinations
* Known allergy to latex when latex products will be in contact with subject
* Pregnant females

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimark, Louisville, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects were recruited from 03.07.2012 - 03.23.2012 from Clinimark LLC, an independent physiology lab.
Pre-assignment Details: Subject distribution requirements (i.e. gender, blood pressure, and arm circumference)were reviewed as part of screening prior to subject enrollment.
Period: Overall Study
Arm/Group | Blood Pressure Reading
Started | 66
Completed | 66
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Blood Pressure Reading
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 45
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 32 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 66
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 125.0 (25.3)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 73 (15.4)
Mean Arterial Pressure (MAP) [Mean (Standard Deviation); unit: mmHg] | 92.7 (17.2)

OUTCOME MEASURES:

1. Primary Outcome: Difference Between the B40 Monitor and Reference Device DINAMAP PRO1000 on NIBP Measurements
Description: The primary endpoints are the difference in systolic, diastolic and mean blood pressure values between the B40 Monitor and PRO1000. The mean of the difference should be no more than 5mmHg and the standard deviation of the difference should be no more than 8mmHg per the AAMI SP-10 standard.
Time Frame: End of each blood pressure reading
Population: 66 subjects were enrolled. 64 subjects contributed data to the study. Subject 058 had a lateral difference of the reference diastolic blood pressure more than 10mmHg, and NIBP data was excluded from final analysis as specified in AAMI SP-10 standard. And Subject 046 had circulation issues and no data was collected.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- B40 and PRO1000 - Systolic BP: Simultaneous blood pressure readings with DINAMAP PRO1000 and B40 monitor; total of 6 successful readings
Arm/Group | B40 and PRO1000 - Systolic BP | B40 and PRO1000 - Diastolic BP | B40 and PRO1000 - MAP
Number analyzed (Participants) | 64 | 64 | 64
mmHg | -1.4 (4.8) | -3.3 (2.6) | -3.7 (4.2)
Statistical Analysis 1: Comparison: B40 and PRO1000 - Systolic BP; A total of no less than 65 subjects are needed for this study. Assuming a mean of no more than 4 mmHg and a standard deviation of no more than 5 mmHg for the difference, this sample size ensures that the percent of subjects with equivalent NIBP is at least 80% with 90% confidence. The difference between the B40 and PRO1000 patient monitors in systolic, diastolic, and mean BP determinations will be compared. A difference of within 10 mmHg is considered equivalent in NIBP; Test type: Non-Inferiority or Equivalence — This study is to show a mean difference of less than 5mmHg and a standard deviation less than 8mmHg for the difference in systolic, diastolic, and mean BP readings taken by B40 and PRO1000 patient monitors; Compare the mean difference with 5mmHg; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.58 to -0.22], Standard Deviation 4.8
Statistical Analysis 2: Comparison: B40 and PRO1000 - Diastolic BP; A total of no less than 65 subjects are needed for this study. Assuming a mean of no more than 4mmHg and a standard deviation of no more than 5mmHg for the difference, this sample size ensures that the percent of subjects with equivalent NIBP is a least 80% with 90% confidence. The difference between the B40 and PRO1000 patient monitors in the systolic, diastolic, and mean BP determinations will be compared. A difference of within 10mmHg is considered equivalent in NIBP; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-3.95 to -2.66], Standard Deviation 2.6
Statistical Analysis 3: Comparison: B40 and PRO1000 - MAP; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-4.73 to -2.67], Standard Deviation 4.2

ADVERSE EVENTS:
Arm/Group | Blood Pressure Reading
Serious Adverse Events (participants affected / at risk) | 0/66
Other Adverse Events (participants affected / at risk) | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor cannot require changes to the PI's disclosure, with the exception of requesting the removal of sponsor's confidential information. The study results themselves are not considered confidential information. Sponsor cannot extend the embargo beyond 60 days unless the PI's disclosure contains patentable subject matter, in which an embargo beyond 60 days may be necessary to allow for the filing of a patent application